CLINICAL TRIAL: NCT06414135
Title: A Dose Ranging Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of Relmacabtagene Autoleucel (Relma-cel) in Patients With Refractory/Progressive Systemic Sclerosis
Brief Title: Relmacabtagene Autoleucel for the Treatment of Systemic Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Liangjing Lu (Other)
Collaborators: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Liangjing Lu, Professor, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029029
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis
Keywords: CAR-T cell therapy; systemic sclerosis; B cell depletion
MeSH Terms: conditions — Scleroderma, Systemic | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relma-cel arm (Experimental): All participants will receive Relma-cel once at different dose levels
  Interventions: Biological: Relma-cel

INTERVENTIONS:
Biological: Relma-cel — All participants will receive Relma-cel once at different dose levels: 25×10^6 CAR+ T cells、50×10^6 CAR+ T cells、75×10^6 CAR+ T cells

SUMMARY:
Relma-cel is a product containing CD19-CAR-transduced T cells. The purpose of this study is to evaluate the safety of Relma-cel at different dose levels in patients with early diffuse systemic sclerosis. Efficacy will be explored too. If enrolled, participants will undergo leukapheresis, lymphodepleting chemotherapy and administration of Relma-cel.

ELIGIBILITY:
Inclusion Criteria:

* voluntary to sign the ICF
* aged between 18-65 years old (inclusive)
* diagnosed with diffuse systemic sclerosis according to 2013 ACR Systemic Sclerosis Classification Criterion
* meet the definitions of refractory/progressive as below:

  1. refractory: non-respondent to or disease recurrence after remission with conventional therapies. Conventional therapies are defined as treated for more than 6 months with low dose steroids (≤ 15 mg prednisone equivalent), cyclophosphamide, antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporin or biologics such as rituximab, belimumab, telitacicept, tocilizumab;
  2. progressive: having below manifestations within 6 months

     1. mRSS increases by >= 3
     2. FVC decreases by > 10% or FVC decreases by > 5% and DLCO decreases by > 15%
* without systemic active infections within 2 weeks of leukapheresis, e.g., infectious pneumonia, tuberculosis
* available vascular access for leukapheresis
* major organ functions:

  1. Renal function: CrCl ≥50 ml/min (Cockcroft/Gault equation)
  2. Bone marrow function: ANC ≥ 1000/uL, absolute lymphocyte count ≥100/uL, Hb ≥90 g/L, Platelet count ≥75 x 10^9/L. Blood transfusion and infusion of growth factors within 7 days of eligibility assessment are not allowed.
  3. Liver function: ALT ≤ 3 x ULN, AST ≤ 3 x ULN, total bilirubin ≤ 2 x ULN (in case of Gilbert syndrome, total bilirubin ≤ 3 x ULN)
  4. Coagulation: INR ≤ 1.5 x ULN, PT ≤1.5 x ULN
  5. Cardiac function: LVEF ≥ 55%
* negative result of serum β-hCG measurement for women of childbearing potential at screening and within 48 hours of the first dose of lymphodepletion
* Female subjects with childbearing potential or male subjects with partners of childbearing potential should adopt medically effective contraception or abstinence from enrollment to 2 years after the end of the study; female subjects with childbearing potential should have a negative serum hCG test within 7 days of enrollment and not in lactation

Exclusion Criteria:

* NYHA class IV
* FVC predicted < 45% or DLCO predicted < 40%
* abnormalities on HRCT not attributable to systemic sclerosis
* history of autologous stem cell transplantation
* with manifestations of renal crisis
* with other autoimmune comorbidities that need systemic treatment
* with a history of severe drug allergy
* with congenital immunoglobulin deficiency
* with malignant tumors, except for nonmelanoma skin cancer, in situ cervical cancer, bladder cancer, breast cancer which has been disease free for more than 2 years
* with psychiatric diseases or severe cognition dysfunctions
* within 5 half-life cycles of the last administration of an investigational product
* pregnant, lactation or plan to be pregnant within one year
* a history of CAR-T therapy or other gene-modified T cell targeted therapies
* other conditions that are not suitable for enrollment of the study in the judgement of the investigator
* the use of any live vaccines against infections within one month of the screening
* with any manifestations of active tuberculosis at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
DLT rate | 28 days
  the incidence of dose-limiting toxicity
Occurrence of AEs and SAEs | 3 months
  frequency and severity of AEs and SAEs

SECONDARY OUTCOMES:
Relma-cel cell numbers and transgene copy numbers and duration in blood | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  Normally Relma-cel number and transgene copy number will gradually decrease to non-measurable as time goes on.
the changes of CD19+ cells and other B cell subsets | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  Theoretically the number of CD19+ cells and other B cell subsets will significantly decreased following Relma-cel administration and gradually increase to normal level as the effect of Relma-cel disappear
the change from baseline in Composite Response Index in Systemic Sclerosis (CRISS) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  Criss is an indicator to evaluate the efficacy of systemic sclerosis therapies. A score greater than or equal to 0.6 means Improvement. A score less than 0.6 means No Improvement.
the change from baseline in Sclerodema Clinical Trial Consortium-Damage Index (SCTC-DI) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  SCTC-DI is a 23-item questionnaire to evaluate the organ damage in patients with systemic sclerosis. The range is between 0-55. The higher the score is, the worse the damage is.
the change from baseline in modified Rodnan Skin Score (mRSS) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  mRSS is an instrument to evaluate cutaneous involvement in patients with systemic sclerosis. The total score ranges from 0 to 51. The higher the score is, the more the cutaneous involvement is.
the change from baseline in pulmonary function (forced vital capacity (FVC) and diffusing capacity of the lungs for carbon monoxide (DLCO)) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  The two items are used to evaluate pulmonary function. Normally both indicators should be greater than 80%.
the change from baseline in cardiac function (left ventricular ejection fraction, LVEF) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  LVEF is an indicator of the heart's ability to eject blood out. The normal range is 50-55%
the change from baseline in high resolution computed tomography (HRCT) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  HRCT is a radiology test of the lungs. In this trial, HRCT will be used to evaluate the lesion size of the lungs, e.g., a lesion could be 10% of the lungs. The greater the percentage is, the worse the lesion is.
the change from baseline in disease activity score -28 (DAS-28) if any joint involvement | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  DAS-28 is a questionnaire to evaluate disease activity in patients with rheumatoid arthritis. 28 joints will be evaluated. Less than 2.6 means the disease is in remission. 2.6-3.2 means a low disease activity. More than 3.2 means active disease needing change in medication. More than 5.1 means very active disease that requires careful monitoring and adjustment to medication
the change from baseline in the levels of inflammation biomarkers including C-reactive protein (CRP), erythropoietin sedimentation rate (ESR) and ferritin | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  CRP, ESR and ferritin are inflammation biomarkers. The normal ranges are different in different labs. Higher values than the upper limit of normal range mean the presence of inflammation.
systemic sclerosis specific antibodies, e.g., anti-scl-70 antibodies, anti-RNA polymerase III antibodies, anti-centrosome antibodies, antinuclear antibody (ANA) | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  Normally all the antibodies are negative in human body. A positive result means abnormalities of immune system.
the change from baseline in skin biopsy pathology, e.g., the number of lymphocytes, the thickness of epiderm | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  In the presence of systemic sclerosis, the increased number of T and B lymphocytes, the thinning of epiderm and the decreased number of sweat gland are expected.
the change from baseline in nailfold capillaroscopy examination, e.g., the capillary density, the diameter of capillaries | 12 months
  nailfold capillaroscopy is a device to observe the capillaries in the nailfold areas. With system sclerosis, the capillary density will diminish and expanded capillary loop may occur
the change from baseline in skin stiffness (measuring the thickness of epiderm and dermis) by skin ultrasound | 12 months
  the thickness of epiderm and dermis will be thinner in the presence of systemic sclerosis.
the change from baseline in health assessment questionnaire -damage index (HAQ-DI) | 12 months
  HAQ-DI, assesses a patient's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in eight categories of functioning which represent a comprehensive set of functional activities - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The stem of each item asks over the past week "Are you able to …" perform a particular task. The patient's responses are made on a scale from zero (no disability) to three (completely disabled). The total score will be 0-3. The higher the score is, the worse the body function is.
the change from baseline in IgG, IgM, IgE, IgA | baseline prior to Relma-cel administration, then through study completion, an average of 2 years after Relma-cel administration
  with Relma-cel administration, IgG, IgM, IgE, IgA will significantly decrease, then graduallly increase as the effect of Relma-cel disappears

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lu, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No